CLINICAL TRIAL: NCT01802554
Title: Reducing CVD Risk in Caregivers: A Brief Behavioral Activation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brent Mausbach, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AG031090 (NIH)
Record Dates: First submitted 2013-02-20; First posted 2013-03-01 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Depressive Symptoms; Inflammation
Keywords: Behavioral Activation; Caregiver; Dementia; Cardiovascular Disease; Alzheimer's Disease; Coagulation
MeSH Terms: conditions — Depression; Inflammation; Dementia; Cardiovascular Diseases; Alzheimer Disease; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pleasant Events Program (PEP) (Experimental): The Pleasant Events Program (PEP) is a Behavioral Activation (BA) treatment for depression. Participants receive 4 weekly sessions of face-to-face therapy (60 minutes each) to increase caregiver participation in pleasurable activities. Two additional phone sessions focus on continued behavioral activation for caregivers as well as problem-solving barriers to activation.
  Interventions: Behavioral: Pleasant Events Program (PEP)
- Information-Support (IS) (Active Comparator): Participants in the Information-Support (IS) control condition were provided with a resource manual consisting of topics commonly covered in support groups or information packets provided by community agencies. Topics included problem-solving and communication skills, cognitive reframing and behavioral management, self-care help, caregiver fact sheets on a range of social and mental health issues, placement information, financial and legal issues, and lists of local organizations and community resources available. Each IS session allowed caregivers to select issue(s) from the resource manual to discuss. The therapist covered the material based on the caregivers' needs. When requested by the caregiver, supportive psychotherapy was also provided.
  Interventions: Behavioral: Information Support (IS)

INTERVENTIONS:
Behavioral: Pleasant Events Program (PEP) — Behavioral Activation Therapy
  Arms: Pleasant Events Program (PEP)
Behavioral: Information Support (IS) — Information-Support (IS) condition consisted of supportive psychotherapy and informational brochures.
  Arms: Information-Support (IS)

SUMMARY:
Cardiovascular disease and depression are some of the most costly illnesses to society, and caring for a loved-one with Alzheimer's disease has been associated with increased risk for both depression and cardiovascular disease. Indeed, depressive symptoms have been linked with elevated plasma concentrations of D-dimer and Interleukin-6 (IL-6), both of which are associated with increased risk for cardiovascular disease (CVD). The present research tests a brief behavioral intervention for reducing both depressive symptoms and CVD biomarkers in Alzheimer caregivers. We hypothesize that caregivers receiving a brief Behavioral Activation (BA) therapy will show greater reductions in depressive symptoms and in CVD biomarkers relative to those randomized to a time-equivalent Information and Support (IS) therapy.

DETAILED DESCRIPTION:
Due to an aging society, the number of people diagnosed with dementia is expected to increase dramatically over the next two decades, with a concomitant rise in the number of family members providing informal care for their loved ones. The stresses associated with this care have been well-documented in the scientific literature, and are noted to be associated with increased risk for psychological and physical morbidity, particularly cardiovascular disease. Indeed, caregiving is associated with elevations in negative affect (e.g., depressive and anxiety symptoms), which in turn is associated with biological indicators that are thought to predict CVD risk (e.g., markers of coagulation and inflammation). The primary goal of this study is to examine the efficacy of a brief Behavioral Activation (BA) Treatment, called the Pleasant Events Program (PEP), for reducing biological CVD risk indicators in a sample of Alzheimer caregivers. We will enroll 100 dementia caregivers and randomly assign them to receive 4-sessions of PEP or 4-sessions of support + information. Our PEP intervention will be conducted in caregivers' homes and will emphasize the importance of monitoring and increasing activities that help individuals make contact with natural reinforcers in their environments, identifying and reducing negative coping responses, and selection and achievement of behavioral goals for healthier living. Caregivers will be assessed for our biological outcomes at baseline, post-treatment, and 1-year to determine intervention efficacy. Given the brief nature of the PEP intervention, the ease with which it can be applied in real-world settings (e.g., community agencies providing services to caregivers), and lack of difficult skills for interventionists and caregivers to acquire, we believe our PEP intervention will be easily transferred to "real-world" settings. If our PEP intervention is efficacious, it may have a considerable impact on both the physical and mental health of caregivers, and will likely have public health implications.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 or older and providing at-home care for a care recipient (CR) with a physician-diagnosis of Alzheimer's disease (AD) or related dementia.

Exclusion Criteria:

* Receiving beta-blocking medications at enrollment
* Receiving treatment with Anticoagulant medications
* Severe hypertension (>200/120 mmHg)
* Diagnosed with a terminal illness with a life expectancy <6 months
* Enrolled in another intervention study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Mausbach, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chattillion EA, Ceglowski J, Roepke SK, von Kanel R, Losada A, Mills PJ, Romero-Moreno R, Grant I, Patterson TL, Mausbach BT. Pleasant events, activity restriction, and blood pressure in dementia caregivers. Health Psychol. 2013 Jul;32(7):793-801. doi: 10.1037/a0029412. Epub 2012 Aug 13. PMID 22888824
- [Background] Mausbach BT, Chattillion E, Roepke SK, Ziegler MG, Milic M, von Kanel R, Dimsdale JE, Mills PJ, Patterson TL, Allison MA, Ancoli-Israel S, Grant I. A longitudinal analysis of the relations among stress, depressive symptoms, leisure satisfaction, and endothelial function in caregivers. Health Psychol. 2012 Jul;31(4):433-40. doi: 10.1037/a0027783. Epub 2012 Apr 9. PMID 22486550
- [Background] Mausbach BT, Roepke SK, Chattillion EA, Harmell AL, Moore R, Romero-Moreno R, Bowie CR, Grant I. Multiple mediators of the relations between caregiving stress and depressive symptoms. Aging Ment Health. 2012;16(1):27-38. doi: 10.1080/13607863.2011.615738. PMID 22224706
- [Background] Chattillion EA, Mausbach BT, Roepke SK, von Kanel R, Mills PJ, Dimsdale JE, Allison M, Ziegler MG, Patterson TL, Ancoli-Israel S, Grant I. Leisure activities, caregiving demands and catecholamine levels in dementia caregivers. Psychol Health. 2012;27(10):1134-49. doi: 10.1080/08870446.2011.637559. Epub 2011 Dec 12. PMID 22149759
- [Background] Mausbach BT, Chattillion EA, Moore RC, Roepke SK, Depp CA, Roesch S. Activity restriction and depression in medical patients and their caregivers: a meta-analysis. Clin Psychol Rev. 2011 Aug;31(6):900-8. doi: 10.1016/j.cpr.2011.04.004. Epub 2011 Apr 28. PMID 21600868
- [Background] Moore RC, Harmell AL, Chattillion E, Ancoli-Israel S, Grant I, Mausbach BT. PEAR model and sleep outcomes in dementia caregivers: influence of activity restriction and pleasant events on sleep disturbances. Int Psychogeriatr. 2011 Nov;23(9):1462-9. doi: 10.1017/S1041610211000512. Epub 2011 Mar 24. PMID 21429282
- [Background] Harmell AL, Chattillion EA, Roepke SK, Mausbach BT. A review of the psychobiology of dementia caregiving: a focus on resilience factors. Curr Psychiatry Rep. 2011 Jun;13(3):219-24. doi: 10.1007/s11920-011-0187-1. PMID 21312008
- [Background] Mausbach BT, Roepke SK, Depp CA, Moore R, Patterson TL, Grant I. Integration of the pleasant events and activity restriction models: development and validation of a "PEAR" model of negative outcomes in Alzheimer's caregivers. Behav Ther. 2011 Mar;42(1):78-88. doi: 10.1016/j.beth.2009.11.006. Epub 2010 Oct 15. PMID 21292054
- [Background] Mausbach BT, Harmell AL, Moore RC, Chattillion EA. Influence of caregiver burden on the association between daily fluctuations in pleasant activities and mood: A daily diary analysis. Behav Res Ther. 2011 Jan;49(1):74-9. doi: 10.1016/j.brat.2010.11.004. Epub 2010 Nov 22. PMID 21130981
- [Background] Mausbach BT, Chattillion EA, Roepke SK, Patterson TL, Grant I. A comparison of psychosocial outcomes in elderly Alzheimer caregivers and noncaregivers. Am J Geriatr Psychiatry. 2013 Jan;21(1):5-13. doi: 10.1016/j.jagp.2012.10.001. Epub 2013 Jan 2. PMID 23290198
- [Result] Moore RC, Chattillion EA, Ceglowski J, Ho J, von Kanel R, Mills PJ, Ziegler MG, Patterson TL, Grant I, Mausbach BT. A randomized clinical trial of Behavioral Activation (BA) therapy for improving psychological and physical health in dementia caregivers: results of the Pleasant Events Program (PEP). Behav Res Ther. 2013 Oct;51(10):623-32. doi: 10.1016/j.brat.2013.07.005. Epub 2013 Jul 19. PMID 23916631

RESULTS

PARTICIPANT FLOW:
Groups:
- Information-Support (IS): Participants in the IS control condition were provided with a resource manual consisting of topics commonly covered in support groups or information packets provided by community agencies. Topics included problem-solving and communication skills, cognitive reframing and behavioral management, self-care help, caregiver fact sheets on a range of social and mental health issues, placement information, financial and legal issues, and lists of local organizations and community resources available. Less structured than the PEP condition, each IS session allowed caregivers to select which issue(s) from the resource manual they would like to discuss, if any, and the therapist covered the material based on the caregivers' needs. When requested by the caregiver, supportive psychotherapy was also provided.
  Information Support (IS) : Supportive Psychotherapy and informational brochures
- Pleasant Events Program (PEP): The Pleasant Events Program (PEP) is a Behavioral Activation (BA) treatment for depression. Participants receive 4 weekly sessions of face-to-face therapy (60 minutes each) to increase caregiver participation in pleasurable activities. Two additional phone sessions focus on continued behavioral activation for caregivers as well as problem-solving barriers to activation.
  Pleasant Events Program (PEP) : Behavioral Activation Therapy
Period: Overall Study
Arm/Group | Information-Support (IS) | Pleasant Events Program (PEP)
Started | 51 | 49
Completed | 43 | 43
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Information Support (IS): Participants in the IS control condition were provided with a resource manual consisting of topics commonly covered in support groups or information packets provided by community agencies. Topics included problem-solving and communication skills, cognitive reframing and behavioral management, self-care help, caregiver fact sheets on a range of social and mental health issues, placement information, financial and legal issues, and lists of local organizations and community resources available. Less structured than the PEP condition, each IS session allowed caregivers to select which issue(s) from the resource manual they would like to discuss, if any, and the therapist covered the material based on the caregivers' needs. When requested by the caregiver, supportive psychotherapy was also provided.
- Total: Total of all reporting groups
Arm/Group | Pleasant Events Program (PEP) | Information Support (IS) | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.86 (7.57) | 71.33 (9.08) | 71.1 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 34 | 74
  Male | 9 | 17 | 26
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Brief Center for Epidemiologic Studies Depression Scale (CESD)
Description: The Brief CESD is a measure of depressive symptoms. The scale's minimum score is 0 and maximum score is 30. Lower scores represent fewer depressive symptoms and thus better outcomes.
Time Frame: Change from Baseline CESD at 8-weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Information-Support (IS): Participants in the IS control condition were provided with a resource manual consisting of topics commonly covered in support groups or information packets provided by community agencies. Topics included problem-solving and communication skills, cognitive reframing and behavioral management, self-care help, caregiver fact sheets on a range of social and mental health issues, placement information, financial and legal issues, and lists of local organizations and community resources available. Less structured than the PEP condition, each IS session allowed caregivers to select which issue(s) from the resource manual they would like to discuss, if any, and the therapist covered the material based on the caregivers' needs. When requested by the caregiver, supportive psychotherapy was also provided.
  Information Support (IS): Supportive Psychotherapy and informational brochures
Arm/Group | Pleasant Events Program (PEP) | Information-Support (IS)
Number analyzed (Participants) | 49 | 51
units on a scale | -3.46 (0.75) | -1.26 (0.74)
Statistical Analysis 1: Comparison: Pleasant Events Program (PEP) vs Information-Support (IS); Test type: Superiority or Other; p = .039, Mixed Models Analysis

2. Primary Outcome: D-dimer
Description: D-dimer is an indicator of fibrin formation and its subsequent lysis and is a useful biomarker representing overall activation of blood coagulation. High concentrations of D-dimer have been linked prospectively to onset of Coronary Heart Disease. Blood was collected by a research nurse in the caregivers' homes through a 22 gauge forearm catheter after a 20 minute rest. Blood for D-dimer was dispensed into polypropylene tubes with 3.8 percent sodium citrate and spun at 1600 g for 10 minutes at room temperature. Obtained plasma was stored at minus 80 degrees Celsius until analyzed. Plasma D-dimer (Asserachrom Stago, Asnieres, France) was determined via high sensitive enzyme-linked immunosorbent assays. Intra- and interassay coefficients of variation were less than 5 percent.
Time Frame: Change from Baseline D-dimer at 8-weeks
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Pleasant Events Program (PEP) | Information-Support (IS)
Number analyzed (Participants) | 49 | 51
ng/ml | -92.22 (56.64) | -61.0 (58.04)
Statistical Analysis 1: Comparison: Pleasant Events Program (PEP) vs Information-Support (IS); Test type: Superiority or Other; p = .701, Mixed Models Analysis

3. Primary Outcome: Interleukin-6 (IL-6)
Description: IL-6 is one of many biomarkers represented in the inflammatory cascade which is initiated during an immune response. Prospectively, increased plasma IL-6 is also associated with future myocardial infarction in healthy men and increasing concentrations of IL-6 have been associated with both nonfatal myocardial infarction and fatal Coronary Heart Disease (CHD) in longitudinal studies of population-based cohorts. Higher concentrations of IL-6 raise CHD risk. Blood was collected by a research nurse in the caregivers' homes through a 22-gauge forearm catheter after a 20 min rest. Blood for IL-6 was dispensed in Ethylenediaminetetraacetic acid (EDTA) tubes and spun at 3000 g for 10 minutes at 4 to 8 degrees Celsius. Obtained plasma was stored at minus 80 degrees Celsius until analyzed. Plasma IL-6 (Meso Scale Discovery, Gaithersburg, MD) was determined via highsensitive enzyme-linked immunosorbent assays. Intra- and interassay coefficients of variation were less than 5 percent.
Time Frame: Change from Baseline IL-6 at 8-weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Pleasant Events Program (PEP) | Information-Support (IS)
Number analyzed (Participants) | 49 | 51
pg/ml | -0.58 (0.66) | 1.33 (0.65)
Statistical Analysis 1: Comparison: Pleasant Events Program (PEP) vs Information-Support (IS); Test type: Superiority or Other; p = .04, Mixed Models Analysis

4. Secondary Outcome: Positive and Negative Affect Schedule
Description: This scales contains ten items assessing Positive Affect. Items included are adjectives, such as "interested," "strong," and "inspired". Participants rated each adjective based on how they felt over the past few weeks using a 5-point scale with responses ranging from 1 (very slightly to not at all) to 5 (extremely). The scale's minimum score is 10 and maximum score is 50. Higher scores represent better outcomes.
Time Frame: Change from Baseline Positive Affect at 8-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pleasant Events Program (PEP) | Information-Support (IS)
Number analyzed (Participants) | 49 | 51
units on a scale | 1.51 (0.82) | 0.23 (0.82)
Statistical Analysis 1: Comparison: Pleasant Events Program (PEP) vs Information-Support (IS); Test type: Superiority or Other; p = .268, Mixed Models Analysis

5. Secondary Outcome: Positive and Negative Affect Schedule
Description: This scales contains ten items assessing Negative Affect. Items included are adjectives, such as "distressed," "ashamed," and Participants rated each adjective based on how they felt over the past few weeks using a 5-point scale with responses ranging from 1 (very slightly to not at all) to 5 (extremely). The scale's minimum score is 10 and maximum score is 50. Lower scores represent better outcomes.
Time Frame: Change from Baseline Negative Affect at 8-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pleasant Events Program (PEP) | Information-Support (IS)
Number analyzed (Participants) | 49 | 51
units on a scale | -3.43 (0.85) | -0.61 (0.85)
Statistical Analysis 1: Comparison: Pleasant Events Program (PEP) vs Information-Support (IS); Test type: Superiority or Other; p = .021, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Pleasant Events Program (PEP) | Information-Support (IS)
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No